CLINICAL TRIAL: NCT05222971
Title: Randomized Open-labeled Phase 2 Study of Maintenance Olaparib With or Without Durvalumab for DDR Gene Mutated Advanced Biliary Tract Cancer Following Platinum-based Chemotherapy
Brief Title: Olaparib With or Without Durvalumab for DDR Gene Mutated Biliary Tract Cancer Following Platinum-based Chemotherapy
Acronym: OPTIMUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMUM
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Biliary Tract Cancer; DNA Damage Repair Deficiency
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — durvalumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olaparib plus durvalumab (Experimental): Olaparib 300 mg twice daily Durvalumab 1,500 mg IV on Day 1
  Every 4 weeks
  Interventions: Drug: Durvalumab; Drug: Olaparib
- Olaparib (Active Comparator): Olaparib 300 mg twice daily
  Every 4 weeks
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1,500 mg IV on Day 1
  Every 4 weeks
  Arms: Olaparib plus durvalumab
Drug: Olaparib — Olaparib 300 mg twice daily
  Every 4 weeks

SUMMARY:
First-line gemcitabine plus cisplatin chemotherapy is the standard first-line treatment for unresectable or metastatic advanced biliary tract cancer and the optimal duration of the treatment is not mentioned in current clinical guidelines. In the pivotal phase 3 ABC-02 trial, patients received up to 6 to 8 cycles of treatment and stopped without maintenance and our retrospective study shows no significant benefit of continuing gemcitabine plus cisplatin beyond 6 to 8 cycles. However, the survival outcomes of patients who completed 6 to 8 cycles of gemcitabine plus cisplatin without progression are dismal with progression-free survival from the last dose of the treatment of median 5.2 months in a prior retrospective study. Indeed, there is an unmet clinical need in terms of maintenance therapy for advanced biliary tract cancer without progression to first-line gemcitabine plus cisplatin chemotherapy.

Durvalumab with/without tremelimumab, anti-CTLA4 inhibitor, showed encouraging results in recently presented study for treatment of advanced biliary tract cancer combination with gemcitabine plus cisplatin. Combination of olaparib and durvalumab showed promising results for metastatic HER-2 negative BRCA mutated breast cancer. For DDR gene mutated advanced biliary tract cancer, olaparib plus durvalumab combination may show synergistic effect with better efficacy than olaparib monotherapy. Both olaparib and durvalumab are relatively well tolerated compared to other cytotoxic chemotherapeutic agents. Olaparib may have some degree of myelosuppression, most patients are expected to well tolerate. Although combination of durvalumab and olaparib may cause additional adverse events, these also might be tolerable, considering that there are no overlapping toxicities between durvalumab and olaparib and the safety data for the combination of durvalumab with olaparib. Considering poor prognosis in patients with advanced biliary tract cancer and lack of maintenance treatment following scheduled first-line GemCis, clinical benefits with maintenance olaparib or olaparib plus durvalumab weigh more than the potential risks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Age 19 years and older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 ~ 1
* Patients must have a life expectancy ≥ 16 weeks.
* Histologically confirmed adenocarcinoma of biliary tract (intrahepatic, extrahepatic cholangiocarcinoma, or gallbladder carcinoma).
* Locally advanced unresectable, recurrence after curative surgery or metastatic disease
* At least 16 weeks of continuous first-line platinum-based chemotherapy for unresectable or metastatic disease
* Somatic or germline mutation of at least one the DNA damage repair gene including ATM, ATR, BAP1, BARD1, BLM, BRCA1, BRCA2, BRIP1, CHEK1, CHEK2, GEN1, FANCA, FANCD2, POLE, MLH1, MSH2, MSH6, MRE11A, NBN, PALB2, PMS2, RAD50, RAD51, RAD51C, RAD51D, and XRCC2 confirmed by targeted exome sequencing
* Measurable disease is not necessarily needed for enrollment.
* No active uncontrolled infection, except chronic viral hepatitis under antiviral therapy.
* Normal organ and bone marrow function measured within 28 days prior to administration of study treatment including haemoglobin ≥10.0 g/dL with no blood transfusion in the past 28 days, platelets ≥ 100 x 109/L, neutrophils ≥ 1.5 x 109/L, creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test ,serum total bilirubin ≤ 1.5 x ULN and alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 x ULN
* No other malignant disease apart from adequately treated non-melanotic skin cancer, curatively treated carcinoma in situ of the uterine cervix, localized prostate or papillary thyroid cancer, or any other cancer where treated with curative intent > 5 years previously without evidence of relapse
* Written, informed consent to the study
* Body weight >30kg
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 6 months.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol or a history of non-compliance
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Obstruction of gastrointestinal tract
* Active gastrointestinal bleeding
* Myocardial infarction within 6 months prior to the study medication, and other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol
* Combined hepatocellular carcinoma/cholangiocarcinoma is excluded.
* ECG abnormalities including mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart), resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with leptomeningeal carcinomatosis or symptomatic uncontrolled brain metastases.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia and vitiligo
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation or double umbilical cord blood transplantation.
* Active or prior documented autoimmune or inflammatory disorders.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Concomitant use of known strong or moderate CYP3A inhibitors/inducers, unless with adequate washout period prior to starting olaparib.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival rate | 6 months
  Time interval between randomization and tumor progression or death of any cause

SECONDARY OUTCOMES:
Overall survival | 1 year
  Time interval between randomization and death of any cauase
Toxicity profile | 6 months
  Any toxicities graded by National Cancer Institute Common Terminology Criteria version 5
Response rates | 6 months
  objective response rates graded by Response Evaluation Criteria in Solid tumor version 1.1
Progression-free survival | 1 year
  Time interval between randomization and tumor progression or death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Study PI will provide IPD to other researchers per request.

REFERENCES:
- [Background] Chae H, Kim D, Yoo C, Kim KP, Jeong JH, Chang HM, Lee SS, Park DH, Song TJ, Hwang S, Kim KH, Song GW, Ahn CS, Lee JH, Hwang DW, Kim SC, Jang SJ, Hong SM, Kim TW, Ryoo BY. Therapeutic relevance of targeted sequencing in management of patients with advanced biliary tract cancer: DNA damage repair gene mutations as a predictive biomarker. Eur J Cancer. 2019 Oct;120:31-39. doi: 10.1016/j.ejca.2019.07.022. Epub 2019 Aug 30. PMID 31476489
- [Background] Domchek SM, Postel-Vinay S, Im SA, Park YH, Delord JP, Italiano A, Alexandre J, You B, Bastian S, Krebs MG, Wang D, Waqar SN, Lanasa M, Rhee J, Gao H, Rocher-Ros V, Jones EV, Gulati S, Coenen-Stass A, Kozarewa I, Lai Z, Angell HK, Opincar L, Herbolsheimer P, Kaufman B. Olaparib and durvalumab in patients with germline BRCA-mutated metastatic breast cancer (MEDIOLA): an open-label, multicentre, phase 1/2, basket study. Lancet Oncol. 2020 Sep;21(9):1155-1164. doi: 10.1016/S1470-2045(20)30324-7. Epub 2020 Aug 6. PMID 32771088
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- [Background] Hyung J, Kim B, Yoo C, Kim KP, Jeong JH, Chang HM, Ryoo BY. Clinical Benefit of Maintenance Therapy for Advanced Biliary Tract Cancer Patients Showing No Progression after First-Line Gemcitabine Plus Cisplatin. Cancer Res Treat. 2019 Jul;51(3):901-909. doi: 10.4143/crt.2018.326. Epub 2018 Oct 4. PMID 30282446
- [Background] Jiao S, Xia W, Yamaguchi H, Wei Y, Chen MK, Hsu JM, Hsu JL, Yu WH, Du Y, Lee HH, Li CW, Chou CK, Lim SO, Chang SS, Litton J, Arun B, Hortobagyi GN, Hung MC. PARP Inhibitor Upregulates PD-L1 Expression and Enhances Cancer-Associated Immunosuppression. Clin Cancer Res. 2017 Jul 15;23(14):3711-3720. doi: 10.1158/1078-0432.CCR-16-3215. Epub 2017 Feb 6. PMID 28167507
- [Background] Kang J, Jeong JH, Hwang HS, Lee SS, Park DH, Oh DW, Song TJ, Kim KH, Hwang S, Hwang DW, Kim SC, Park JH, Hong SM, Kim KP, Ryoo BY, Yoo C. Efficacy and Safety of Pembrolizumab in Patients with Refractory Advanced Biliary Tract Cancer: Tumor Proportion Score as a Potential Biomarker for Response. Cancer Res Treat. 2020 Apr;52(2):594-603. doi: 10.4143/crt.2019.493. Epub 2019 Dec 18. PMID 32019287
- [Background] Teo MY, Seier K, Ostrovnaya I, Regazzi AM, Kania BE, Moran MM, Cipolla CK, Bluth MJ, Chaim J, Al-Ahmadie H, Snyder A, Carlo MI, Solit DB, Berger MF, Funt S, Wolchok JD, Iyer G, Bajorin DF, Callahan MK, Rosenberg JE. Alterations in DNA Damage Response and Repair Genes as Potential Marker of Clinical Benefit From PD-1/PD-L1 Blockade in Advanced Urothelial Cancers. J Clin Oncol. 2018 Jun 10;36(17):1685-1694. doi: 10.1200/JCO.2017.75.7740. Epub 2018 Feb 28. PMID 29489427
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404